CLINICAL TRIAL: NCT01232140
Title: CRP-guided Antibiotic Treatment in Patients Hospitalized With Acute Exacerbations of COPD Patients. A Randomized Controlled Intervention Trial.
Brief Title: CRP-guided Antibiotic Treatment in COPD Exacerbations Admitted to the Hospital
Acronym: CATCH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical Center Alkmaar (Other)
Responsible Party: Principal Investigator, W.G.Boersma, PhD, Medical Center Alkmaar
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CATCH study; AECOPD (Other Grant/Funding Number: Foreest Medical School Medical Center Alkmaar)
Record Dates: First submitted 2010-11-01; First posted 2010-11-02 (Estimated); Last update posted 2012-03-22 (Estimated); Status verified 2012-03

CONDITIONS: COPD; Exacerbation; Bronchitis; Sputum; C-Reactive Protein
Keywords: COPD; exacerbation; antibiotic treatment; CRP; sputum; inflammation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CRP-guided antibiotic treatment (Experimental): If CRP> 50 mg/l a patient receive antibiotic treatment, whereas in those patients with CRP =< 50 mg/l antibiotic treatment is withheld.
  Interventions: Other: CRP-guided antibiotic treatment
- GOLD strategy-antibiotic treatment (Other): According to the GOLD strategy a patient with an AECOPD should prescribed antibiotic treatment if a patient has symptoms of increased dyspnea, increased sputum production and change of sputum color. Two of these three criteria should be present, however change in sputum production is obligatory.
  Interventions: Other: CRP-guided antibiotic treatment

INTERVENTIONS:
Other: CRP-guided antibiotic treatment — If CRP> 50 mg/l patients with AECOPD receive antibiotic treatment, whereas in those patients with CRP =< 50 mg/l antibiotic treatment are withheld. This will be compared to the regular antibiotic treatment that has been advised by the GOLD strategy

SUMMARY:
Rationale: Acute exacerbations are key events in chronic obstructive pulmonary disease (COPD), resulting in poorer quality of life. Causes include irritants, viruses and bacterial pathogens. These exacerbations are often treated with a combination of corticosteroids, bronchodilators and antibiotics, but the benefit of antibiotic therapy remains controversial. Several trials studying antibiotic treatment in AECOPD showed conflicting data, with several large studies failing to demonstrate superiority of antibiotic therapy over placebo. Other trials indicated that antibiotic therapy is effective in patients who have at least two of the following symptoms: increased dyspnoea, increased sputum volume and increased sputum purulence. Ever since sputum purulence has been used as a predictive marker in AECOPD, a strategy that has been integrated in the GOLD guideline for treatment of AECOPD. However, the color of sputum reported by patients is not always reliable and inspection of sputum is not always possible. Several serum biomarkers such as C-reactive protein (CRP) and procalcitonin (PCT) are now available. In a recent trial of doxycycline in addition to systemic corticosteroids for patients hospitalized with AECOPD we found that CRP might be valuable as a marker predictive of response to antibiotic treatment in AECOPD.

DETAILED DESCRIPTION:
Objective: CRP-guided antibiotic therapy will be compared with standard antibiotic therapy in AECOPD. Our aim is that CRP guided therapy will lead to 20% reduction in antibiotic consumption.

Study design: randomized controlled intervention trial Study population: Hospitalised COPD patients with acute exacerbation. Intervention (if applicable): Patients with type 1 and 2 exacerbation will be assigned to either CRP guided therapy or antibiotic therapy according to GOLD guidelines.

Main study parameters/endpoints: The main endpoint of the study is the reduction in antibiotic consumption. Furthermore, the real incidence of infiltrates in AECOPD with fever will be studied. As secondary outcome the objectives length of hospitalization, time to treatment failure within 30-days and time to next exacerbation will be assessed. The relation between the level of biomarkers the presence of infiltrates on the HRCT will be investigated.

Subjective improvement in symptoms will be measured by symptoms (VAS-LRTI) and quality of life will be assessed by St George's Respiratory Questionnaire. Finally, adverse effects of the antibiotic treatment will be recorded.

In order to observe a significant difference of antibiotic consumption, 60% in standard antibiotic group and 40% in CRP guided antibiotic group, with a power of 0.8, a total of 110 patients have to be assigned by randomisation to each group.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Patients in both treatment arms will receive a non-experimental treatment. Both treatment options are recognized as part of standard care. The burden associated with participation is limited to a total of 3 visits to the hospital and phone call for data assessment at regular follow-up. There are no specific risks involved in participating. Less adverse effects may be beneficially for the patient.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 or over. No upper age limit will be employed.
* Written informed consent obtained.
* AECOPD according to the GOLD guideline. An exacerbation of COPD is defined as an event in the natural course of the disease characterized by a change in the patient's baseline dyspnoea, cough, and/or sputum that is beyond normal day-to-day variations, is acute in onset, and may warrant a change in regular medication in a patient with underlying COPD.
* Criteria for hospital admission according to the GOLD: marked increase in symptoms (i.e. resting dyspnoea), severe underlying COPD, onset of new physical signs (cyanosis, edema), failure to respond to initial medical management, significant co morbidities, frequent exacerbations, newly occurring arrhythmias, diagnostic uncertainty.
* Former of current smoker with a minimum smoking history of 10 pack years.
* Patients have to be capable of ingesting oral medication.
* Patients have to be mentally capable of participating in the study (able to complete questionnaires and perform lung function tests).
* Life expectancy ≥ 30 days.

Exclusion Criteria:

* Pregnant or lactating women, or women of childbearing age not using an acceptable method of contraception.
* Pretreatment with corticosteroids (cumulative dose >210 mg) for the present exacerbation.
* Progression or new radiographic abnormalities on the chest X-ray or CT scan compatible with pneumonia.
* bronchiectasis (HRCT confirmed).
* Cystic fibrosis.
* Tuberculosis.
* Immunodeficiency disorders such as AIDS, humoral immune defect, ciliary dysfunction etc., and the use of immunosuppressive drugs (>30 mg prednisolone/day maintenance dose or equivalent for more than 4 weeks).
* Recent or unresolved lung malignancy.
* Other disease likely to require antibiotic therapy, such as recurrent sinusitis or urinary tract infection.
* Significant gastrointestinal or other conditions that may affect study drug absorption.
* Class III or IV congestive heart failure or stroke.
* Newly diagnosed pulmonary embolism

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2011-07; Primary Completion 2013-03 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Number of patients treated with antibiotics during hospital stay | 10 days
  Sputum purulence has been used as a predictive marker in AECOPD.However, the color of sputum reported by patients is not always reliable and inspection of sputum is not always possible. Serum biomarker such as C-reactive protein (CRP) represents systemic inflammation.In the present study, we will compare CRP guided antibiotic treatment versus treatment according to GOLD strategy. Our hyposthesis is that CRP-guided therapy results in lower number of antibiotic prescriptions

SECONDARY OUTCOMES:
Time to treatment failure within 30-days | 30 days
  Treatment failure within 30 days after hospital admission will be compared
Length of stay | 30 days
  Length of hospital stay for the exacerbation
Time to next exacerbation | 1 year
  Time to the next exacerbation with a follow-up period of one year
Symptom scores (VAS-LRTI, George's Respiratory Questionnaire) | 30 days
  Symptom score (VAS-LRTI) and Quality of life (George's Respiratory Questionnaire) will be measured at onset and recovery.
Adverse events | 30 days
  Adverse events of antibiotic treatment are recorded during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: W.G. Boersma, PHD,MD, Study Director — Medical Centre Alkmaar
Locations (1):
- W.G.Boersma, Alkmaar, North Holland, Netherlands

REFERENCES:
- [Result] Daniels JM, Snijders D, de Graaff CS, Vlaspolder F, Jansen HM, Boersma WG. Antibiotics in addition to systemic corticosteroids for acute exacerbations of chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2010 Jan 15;181(2):150-7. doi: 10.1164/rccm.200906-0837OC. Epub 2009 Oct 29. PMID 19875685
- [Derived] Prins HJ, Duijkers R, Daniels JMA, van der Molen T, van der Werf TS, Boersma W. COPD-Lower Respiratory Tract Infection Visual Analogue Score (c-LRTI-VAS) validation in stable and exacerbated patients with COPD. BMJ Open Respir Res. 2021 Feb;8(1):e000761. doi: 10.1136/bmjresp-2020-000761. PMID 33593795
- [Derived] Prins HJ, Duijkers R, Lutter R, Daniels JM, van der Valk P, Schoorl M, Kerstjens HA, van der Werf TS, Boersma WG. Blood eosinophilia as a marker of early and late treatment failure in severe acute exacerbations of COPD. Respir Med. 2017 Oct;131:118-124. doi: 10.1016/j.rmed.2017.07.064. Epub 2017 Aug 1. PMID 28947018